CLINICAL TRIAL: NCT05514951
Title: Study of the Prevalence of Iron Deficiency in Elderly Patient in Hospital Environment
Acronym: CARENFERPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vifor Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A00787-36
Record Dates: First submitted 2022-08-22; First posted 2022-08-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Iron-deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sampling (Experimental): Blood sampling
  Interventions: Diagnostic Test: Blood sampling

INTERVENTIONS:
Diagnostic Test: Blood sampling — Blood sampling

SUMMARY:
Iron deficiency is defined by insufficient tissue iron stores and anemia is the ultimate stage of iron deficiency. Anemia should never be neglected in an elderly subject because it is associated with an increase in mortality, but also with a increased morbidity in terms of complications

Apart from anemia, iron deficiency is common and constitutes a factor of poor prognosis in diseases chronic, all pathologies very frequently found in the elderly. It is the origin of the deterioration in the general condition of patients, their re-hospitalization or even the progression of their pathology.

In this context where elderly patients also present a certain number of comorbidities including the pathologies mentioned previously, it is important to better diagnose the deficiency martial in the elderly patient.

DETAILED DESCRIPTION:
Iron deficiency (MD) is defined by insufficient tissue iron stores. Since iron is essential for the synthesis of hemoglobin, when the iron deficiency no longer makes it possible to maintain a sufficient level of erythropoiesis, anemia appears: it is the ultimate stage of iron deficiency.

Anemia is the most common haematological pathology encountered in geriatric practice. Its prevalence, in population generally ambulatory, is between 10 and 15% after the age of 65 and is greater than 20% beyond the age of 85.

Anemia should never be neglected in an elderly subject because it is associated with an increase in mortality, but also with a increased morbidity in terms of complications heart disease, cognitive decline, frailty, hospitalizations, and impairment of quality of life. About a third of anemias elderly person is attributable to a deficiency in vitamin B9 or B12 or an iron deficiency.

Apart from anemia, iron deficiency is common and constitutes a factor of poor prognosis in diseases chronic such as heart failure, kidney failure chronic or cancer, all pathologies very frequently found in the elderly. It is the origin of the deterioration in the general condition of patients, their re-hospitalization or even the progression of their pathology.

In this context where elderly patients also present a certain number of comorbidities including the pathologies mentioned previously, it is important to better diagnose the deficiency martial in the elderly patient.

This diagnosis is all the more important because, depending on the chronic pathology, data from the literature have shown that correcting the iron deficiency brings benefits to the patient by reducing the risk of recurrence of anemia, the prescription of erythropoietin and the use of transfusion for patients in oncology, gastroenterology and nephrology

ELIGIBILITY:
Inclusion Criteria:

* Any patient hospitalized in a geriatric unit (short geriatric stay, SSR) or seen on an outpatient basis (hospitalization day, consultation)
* Affiliated patient or beneficiary of a social healthcare system
* Patient having given written consent

Exclusion Criteria:

* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by court order or administration

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 888 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients diagnosed with iron deficiency on inclusion | Day 1
  The diagnosis of iron deficiency will be made from the measurements of the ferritinemia and CST: Ferritinemia < 100 µg/L and/or CST < 20%

CONTACTS AND LOCATIONS:
Locations (16):
- France (16):
  - Chu Angers, Angers
  - CH de Bayonne, Bayonne
  - Ch De Calais, Calais
  - CH Chambéry, Chambéry
  - CHSF, Corbeil-Essonnes
  - Ch de Dunkerque, Dunkirk
  - Hôpital Gériatrique Les Bateliers Chu Lille, Lille
  - Chu De Nantes, Hôpital Bellier, Nantes
  - CHU de NICE-hopital CIMIEZ, Nice
  - Hopital Saint Antoine, Paris
  - CH de Pau, Pau
  - CHU de Poitiers, Poitiers
  - HUS - Hôpitaux Universitaires de Starsbourg, Strasbourg
  - Hôpital Bretonneau, Tours
  - Chu Nancy, Vandœuvre-lès-Nancy
  - HCL, Villeurbanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fougere B, Puisieux F, Chevalet P, Annweiler C, Michel E, Joly L, Blanc F, Azouzi AE, Desre-Follet V, Cacoub P; CARENFER PA study group*. Prevalence of iron deficiency in patients admitted to a geriatric unit: a multicenter cross-sectional study. BMC Geriatr. 2024 Jan 30;24(1):112. doi: 10.1186/s12877-024-04719-6. PMID 38287253